CLINICAL TRIAL: NCT03760562
Title: The Risk of Hypertension Associated With Oral Glucocorticoids in Chronic Inflammatory Diseases in England.
Brief Title: The Risk of Hypertension Associated With Oral Glucocorticoids in Chronic Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Mar Pujades Rodriguez, Principal Investigator, University of Leeds
Other Study IDs: 16_146H
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Glucocorticoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Glucocorticoids — Oral Glucocorticoids.

SUMMARY:
Glucocorticoids are widely used for the treatment of chronic inflammatory diseases. In 2008, it was estimated that 0.8% of the United Kingdom adult population had used long-term (≥ 3 months) glucocorticoids, rising to 3% in women aged over 80 years.

The aim of the project is to investigate the dose-response estimates of risk of high blood pressure associated with oral glucocorticoids.

DETAILED DESCRIPTION:
Hypertension is a chronic condition which affects 1 in 5 of the world adult population. The cause of hypertension is unknown in about 95% of patients, whilst 5% are secondary to underlying adrenal disorders or other identifiable causes.

Glucocorticoids are widely used for the treatment of chronic inflammatory diseases. In 2008, it was estimated that 0.8% of the UK adult population had used long-term (≥ 3 months) glucocorticoids, rising to 3% in women aged over 80 years. Glucocorticoids are effective in controlling underlying chronic inflammatory disease in majority of cases. However, their continuous use can result in a variety of complications, including hypertension.Although it is acknowledged that excess cortisol is a leading cause of hypertension, the role of exogenous glucocorticoids is less known.

The aim of the project is to investigate the dose-response estimates of risk of high blood pressure associated with oral glucocorticoids.

This is a retrospective cohort study of people diagnosed with at least one of six chronic inflammatory diseases (polymyalgia rheumatica, giant cell arteritis, systemic lupus erythematosus, rheumatoid arthritis, vasculitis and inflammatory bowel disease). This study will be based on the analysis of existing primary care health records routinely collected, linked to hospital and mortality data.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old or over
* Registered in a participating general practice 1 year or more during the study period
* Minimum of 1 year prior to study entry meeting CPRD data quality
* Diagnosed with at least one of the 6 chronic inflammatory diseases

Exclusion Criteria:

* Patients aged under 18 years during the study period
* Registered in general practices that did not consent to data linkage

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients registered in Clinical Practice Research Datalink (CPRD) who were eligible for data linkage and had been diagnosed with at least one of six chronic inflammatory diseases (inflammatory bowel diseases, systemic lupus erythematosus, polymyalgia rheumatica, giant cell arteritis, rheumatoid arthritis, and vasculitis) in the period between 1st Jan 1998 and 15th March 2017.
Sampling Method: Non-Probability Sample
Enrollment: 111804 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Glucocorticoid-related hypertension | 18 years
  Number of patients with incident hypertension

REFERENCES:
- [Derived] Mebrahtu TF, Morgan AW, West RM, Stewart PM, Pujades-Rodriguez M. Oral glucocorticoids and incidence of hypertension in people with chronic inflammatory diseases: a population-based cohort study. CMAJ. 2020 Mar 23;192(12):E295-E301. doi: 10.1503/cmaj.191012. PMID 32392512